CLINICAL TRIAL: NCT01259544
Title: BreathID® Test: A Non-invasive Modality to Detect Pancreatic Exocrine Insufficiency
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Meridian Bioscience, Inc. (Industry)
Collaborators: Virginia Commonwealth University (Other); Asian Institute of Gastroenterology, Hyderabad, India (Unknown)
Responsible Party: Bimaljit S Sandhu, M.D, Virginia Commonwealth University Medical Center
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Diagnostic
Other Study IDs: CP-EX-110
Record Dates: First submitted 2010-12-12; First posted 2010-12-14 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Chronic Pancreatitis; Healthy Volunteers
Keywords: CP-Chronic Pancreatitis; DPT-Di peptide breath test; ePFT- Endoscopic pancreatic function test
MeSH Terms: conditions — Pancreatitis, Chronic | interventions — benzoyl-tyrosyl-alanine

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Di -petide breath tests and ePFT secretin induced (Active Comparator): Di peptide breath tests will be performed on subjects with known chronic pancreatitis
  Interventions: Drug: benzoyl-L-tyrosyl-[1-13C]alanine (Bz-Tyr-Ala)
- c13 di peptide breath tests (Active Comparator): Healthy volunteers to compare breath tests results to subjects with chronic pancreatitis
  Interventions: Drug: benzoyl-L-tyrosyl-[1-13C]alanine (Bz-Tyr-Ala)

INTERVENTIONS:
Drug: benzoyl-L-tyrosyl-[1-13C]alanine (Bz-Tyr-Ala) — 300 mg of powder form dissolved in one cup of tap water prior to breath test
  Arms: Di -petide breath tests and ePFT secretin induced
Drug: benzoyl-L-tyrosyl-[1-13C]alanine (Bz-Tyr-Ala) — 300 mg of 13 C di peptide in single dose powder form dissolved in one cup of tap water.
  Arms: c13 di peptide breath tests

SUMMARY:
13C breath di-peptide tests are an effective non-invasive tool to detect pancreatic exocrine function in patients with Chronic Pancreatitis.

DETAILED DESCRIPTION:
The aim of the study is to assess the pancreatic exocrine insufficiency using a 13C labeled di-peptide breath tests in patients with chronic pancreatitis(CP) and show correlation with secretin stimulated endoscopic Pancreatic Function Test (ePFT). Furthermore, a second purpose is to assess the ability to differentiate between non patients with chronic pancreatitis and those without. Approximately 30 subjects will be tested with both methods within two weeks of each other.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with chronic pancreatitis who meet at least one of the following criteria:

   * Adult men or women >18 years of age.
   * Endoscopic retrograde cholangiopancreatography (ERCP), magnetic resonance cholangiopancreatography (MRCP), or endoscopic ultrasound demonstrating ductal changes consistent with chronic pancreatitis
   * Abnormal secretin pancreatic function test with a peak bicarbonate concentration <80 mEq/L
   * Presence of pathogenomic pancreatic calcifications
   * Pathology proven chronic pancreatitis on surgical specimens
2. Females of childbearing potential must be willing to use birth control (IUD, oral, transdermal, parenteral contraceptives, or abstinence)
3. Patients who can fast for at least 8 hours
4. Able to perform the testing and procedures required for the study, as judged by the investigator
5. Willing and able to provide written informed consent

Exclusion Criteria:

* Failure to obtain consent
* Patients with liver cirrhosis
* Any co-morbid condition with expected survival < 1 year
* History of extensive bowel resection, multiple abdominal surgeries
* Women who are pregnant, breastfeeding, or of childbearing potential and not willing to use methods of birth control
* Uncontrolled diabetes
* Patients currently receiving total parenteral nutrition (TPN)
* Recipients of an organ transplant
* Patients who have consumed >20cc of alcohol or have taken acetaminophen in the past 24 hours
* History of chronic obstructive pulmonary disease or symptomatic bronchial asthma
* Patients taking drugs that can interfere with 13C di-peptide metabolization

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2009-01; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
To assess the pancreatic exocrine insufficiency using a 13C labeled di-peptide breath tests in patients with chronic pancreatitis(CP) and show correlation with secretin stimulated endoscopic Pancreatic Function Test (ePFT). | 1 hour
  This breath test substrate is new and is hypothesized, based on preliminary studies, that it may be the answer to a much needed non-invasive pancreatic function test. At first stage, it will be compared to the current invasive gold standard: secretin induced ePFT.

SECONDARY OUTCOMES:
To assess the ability to differentiate between non patients with chronic pancreatitis and those without. | 1 hour
  In order to establish the efficacy of this test, it is necessary to confirm that a difference is observed between healthy and non- healthy subjects

CONTACTS AND LOCATIONS:
Locations (1):
- Asian Institute of Gastroenterology, Hyderabad, India, Somājigūda, Hyderabad, India